CLINICAL TRIAL: NCT06591611
Title: Effect of PEEK and Co-Cr Framework Reinforcement on Marginal Bone Loss Around Implants Supporting a Fixed All-on-four Prosthesis in Completely Edentulous Mandibles. A Randomized Controlled Clinical Trial
Brief Title: Effect of PEEK and Co-Cr Framework Reinforcement on Marginal Bone Loss Around Implants Supporting a Fixed All-on-four Prosthesis in Completely Edentulous Mandibles. A Randomized Controlled Clinial Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, shereen ismail, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21223
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: All on Four, Marginal Bone Loss, PEEK
MeSH Terms: interventions — Dental Prosthesis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-Cr reinforced fixed all-on-four prosthesis (Active Comparator)
  Interventions: Other: PEEK reinforced fixed all-on-four prosthesis
- PEEK reinforced fixed all-on-four prosthesis (Experimental)
  Interventions: Other: PEEK reinforced fixed all-on-four prosthesis

INTERVENTIONS:
Other: PEEK reinforced fixed all-on-four prosthesis — Fabricating a fixed prosthesis for patients with completely edentulous mandibles reinforced with PEEK
  Other Names: Dental Prosthesis

SUMMARY:
A fixed all-on-four prosthesis will be fabricated for the mandibular arch for each patient and the marginal bone loss will be evaluated at baseline, 3,6,9 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patient with old satisfactory maxillary and mandibular dentures requiring an implant supported restoration
* Implant sites must allow for implant placement
* Patients with no systemic conditions that may interfere with implant placement

Exclusion Criteria:

* General contraindications for implant surgery( Poor oral hygiene- diabetes- pregnancy or nursing- drug abusers)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss | 12 months
  marginal bone loss around each implant

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No